CLINICAL TRIAL: NCT05124639
Title: A Pragmatic Randomized Controlled Trial of a Group Self-management Support Program Versus Treatment-as-usual for Anxiety Disorders
Brief Title: Clinical Trial of a Group Self-management Support Program for Anxiety Disorders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Relief (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PJT-169163
Record Dates: First submitted 2021-10-27; First posted 2021-11-18 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Panic Disorder; Agoraphobia; Social Anxiety Disorder; Generalized Anxiety Disorder
Keywords: Panic Disorder; Agoraphobia; Social Anxiety Disorder; Generalized Anxiety Disorder; Anxiety disorders; Self-management support
MeSH Terms: conditions — Panic Disorder; Agoraphobia; Phobia, Social; Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group self-management support (Experimental): Group self-management support program for anxiety disorders developped by Relief (https://myrelief.ca/).
  Interventions: Behavioral: Group self-management support program for anxiety disorders
- Treatment-as-usual (No Intervention): Treatment-as-usual and a delayed intervention (if desired by participants) after the 12-month follow up

INTERVENTIONS:
Behavioral: Group self-management support program for anxiety disorders — The group SMS manualized program for anxiety disorders (https://monrelief.ca) aims at improving self-management capabilities through weekly 2.5-hours sessions with 10-15 patients over a 10-week period.This trial will focus solely on the virtual format of the program. The SMS program covers the following themes: getting to know your anxiety; building self-awareness; reconsidering your lifestyle habits; adopting a problem-solving method; avoidance and exposure; acceptance and committed action; seeing things differently; managing your emotions; receiving support from others; and consolidating your toolkit.
  Other Names: SMS+TAU
  Arms: Group self-management support

SUMMARY:
Background. Self-management support is a complementary approach to treatment that aims to educate participants on the nature of anxiety and to improve their strategies to manage symptoms and well-being, thus presenting the potential to enhance recovery, improve outcomes, reduce recurrence rates and lower health care costs. There is limited evidence to support the effectiveness of group self-management support for anxiety disorders in community-based care.

Objectives. This study aims at examining the effectiveness of a virtual group self-management support program (SMS) for anxiety disorders as an add-on to treatment-as-usual (TAU) in community-based care settings. We will also assess the incremental cost/effectiveness ratio and the implementability of the intervention.

Methods. The trial is a pragmatic randomized controlled trial with a pre-treatment, post-treatment (4-month post-randomization), and follow-ups at 8, 12 and 24-months. Intervention. The experimental condition will consist of a 10-week SMS program for anxiety disorders in addition to TAU. The control condition will receive TAU without restrictions for anxiety disorders. Inclusion criteria will comprise being 18 years old or older, French-speaking, and presenting symptoms of anxiety disorders based on self-reported validated assessment scales. Patients will be recruited in the province of Quebec (Canada). Outcome measures: The primary outcome measure is the Beck Anxiety Inventory (BAI). The secondary outcome measures include self-reported instruments for anxiety and depressive symptoms, recovery, self-management, quality of life, and service utilisation. Statistical analysis: Intention-to-treat analysis. A mixed effects regression model will be used to account for between and within-subject variations in the analysis of the longitudinal effects of the intervention.

Expected outcomes. The rigorous evaluation of the SMS intervention in the real world will provide information to decision makers, health care managers, clinicians and patients regarding the added value of group SMS for patients with anxiety disorders. Widespread implementation of this intervention could lead to more efficient mental health care services, to better long-term outcomes and to a significant reduction in the extensive social and economic burden of anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* (1) aged 18 and over,
* (2) fluent in spoken and written French,
* (3) presence of symptoms of anxiety disorders based on self-reported validated assessment scales and semi-structured assessment interview,
* (4) access to a computer or tablet connected to the internet with microphone and video camera

Exclusion Criteria:

* (1) previous enrolment in the SMS intervention provided by Relief
* (2) active suicidal intentions,
* (3) severe depressive symptoms,
* (4) active substance-related and addictive disorder,
* (5) cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Anxiety Inventory (BAI) | Baseline and post-treatment (4-month post-randomization)

SECONDARY OUTCOMES:
Change in Beck Anxiety Inventory | Baseline, post-treatment, and 8-month, 12-month, 24-month post-randomization follow-ups
Change in Generalised Anxiety Disorder-7 | Baseline, post-treatment, and 8-month, 12-month, 24-month post-randomization follow-ups
Change in Patient Health Questionnaire-9 | Baseline, post-treatment,12-month and 24-month post-randomization follow-ups
Change in Recovery Assessment Scale - Revised | Baseline, post-treatment,12-month and 24-month post-randomization follow-ups
Change in Mental Health Self-Management Questionnaire | Baseline, post-treatment,12-month and 24-month post-randomization follow-ups
Change in Assessment of Quality of Life - 6 Dimensions | Baseline, post-treatment, and 8-month, 12-month, 24-month post-randomization follow-ups
Change in Health care use and indirect costs | Baseline, post-treatment, and 8-month, 12-month, 24-month post-randomization follow-ups
  Health care costs for other mental health consultations (e.g. type of professional, duration, costs), psychotherapy experience (including CBT) and psychotropic medication.
Change in Administrative databases records | Starting 12 months prior to participant enrolment up to the 24-month post-randomization follow-up
  Data will be obtained from provincial administrative databases for medical and biopsychosocial services, hospitalization's registry, and medication data.

OTHER OUTCOMES:
Gross Cohesion Scale | During the 10-week SMS program, after sessions 3 and 8 (for experimental arm participants)
Working Alliance Inventory | During the 10-week SMS program, after sessions 3 and 8 (for experimental arm participants)

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Roberge, Ph.D., Principal Investigator — Université de Sherbrooke; Janie Houle, Ph.D., Principal Investigator — Université du Québec a Montréal
Locations (1):
- Université de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available on request from the nominated principal investigator [PR]. The data will not be publicly available due to ethics approval restrictions.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Roberge P, Houle J, Provost JR, Coulombe S, Beaudin A, Bower P, Lemyre FC, Drapeau M, Drouin MS, Hudon C, Provencher MD, Vasiliadis HM. A pragmatic randomized controlled trial of a group self-management support program versus treatment-as-usual for anxiety disorders: study protocol. BMC Psychiatry. 2022 Feb 21;22(1):135. doi: 10.1186/s12888-021-03675-4. PMID 35189848
- See also: Developper of the SMS-A program — https://relief.ca/relief-1/home
- See also: Nominated principal investigator's [PR] laboratory website. — https://proberge.recherche.usherbrooke.ca
- See also: Published study protocol in BMC Psychiatry — https://doi.org/10.1186/s12888-021-03675-4